CLINICAL TRIAL: NCT01291875
Title: Periodontal Treatment and Metabolic Control in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Chairman of Periodontics Department, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 127/2009
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus; Periodontal Disease
Keywords: Type 2 Diabetes mellitus; Periodontal Disease; metabolic control; periodontal treatment; inflammatory markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive periodontal treatment (Experimental)
  Interventions: Procedure: non-surgical periodontal treatment
- Supragingival biofilm control (Active Comparator)
  Interventions: Procedure: Supragingival biofilm control

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — Patients in this group will receive a non surgical periodontal therapy: scaling and root planing of the root surfaces under local analgesia (depending on the severity in one session or two sessions within 2 days). Any tooth that from the baseline examination is defined as hopeless or irrationale to treat will be extracted. After to 2 months re-assessment presenting at least one periodontal site with pocket depth of 6 mm will have additional corrective periodontal therapy.
  Arms: Intensive periodontal treatment
Procedure: Supragingival biofilm control — Control group patients will receive a standard cycle of supra-gingival mechanical instrumentation and polishing in one appointment performed as appropriate by a single clinician using a combination of hand and machine driven (piezoelectric) instrumentation.
  Arms: Supragingival biofilm control

SUMMARY:
The studies that correlate periodontal disease (PD) and diabetes mellitus (DM) suggest that individuals with poor glycemic control are at increased risk for developing infections. Despite being controlled for other important risk factors, diabetic patients are three times more likely to develop PD, and therefore, periodontitis has been proposed as the sixth complication of DM.

Besides the effect of diabetes on DP, the reverse has also been studied over the past 15 years, through the idea that chronic and acute infections can directly affect the tissue resistance to insulin. Recent studies have provided evidence that controlling periodontal infection has an impact on improvement of glycemic control in diabetes mellitus patients. The vascularity of the inflamed periodontal tissue serves as a gateway to inflammatory mediators, pathogenic bacteria and their products into the bloodstream. Some researchers have suggested that periodontal treatment in type 2 diabetes mellitus (DMT2) patients, results in beneficial effect on the level of glycemic control. However, there is no conclusive evidence to support this hypothesis.

This research project aims to determinate the impact of periodontal therapy on metabolic control in DMT2 individuals, and determinate the possible association between periodontal disease and DMT2. For the HbA1c outcome this clinical trial had a sample size calculation estimated at 120 patients. For the inflammatory serum markers this study had a sample size estimated at 22 individuals. Blood samples will be collected for evaluation of Hba1c and inflammatory serum markers. This data will highlight the possible role of periodontal therapy on DMT2 metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged over 30 years old
* Subject diagnosed with T2DM
* Subject consenting to the study
* Subject with signs of severe periodontitis (at least 50 periodontal pockets, PPD > 4mm and Bleeding on Probing)

Exclusion Criteria:

* Pregnancy - Lactation
* Subject is on chronic treatment (i.e., two weeks or more) with specific medications known to affect periodontal status (phenytoin or cyclosporine) within one month of baseline visit
* Subject with known HIV or Hepatitis (B, C)
* Subjects with uncontrolled systemic diseases (cardiovascular diseases including hypertension, liver, pulmonary diseases, end stage renal failure) and/or neoplasm
* Subjects not capable to provide informed consent
* Subjects on chronic antibiotic therapy or who require antibiotic coverage for periodontal procedures

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c and serum inflammatory markers of inflammation after periodontal intervention | It will be assessed 2, 6 and 12 months after periodontal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry - University of São Paulo, São Paulo, Brazil